CLINICAL TRIAL: NCT05980546
Title: A Randomized Controlled Trial of Ultrasound Guided Knee Genicular Nerve Block and Anterior Femoral Cutaneous Nerve Block for Primary Total Knee Arthroplasty
Brief Title: Genicular and Anterior Femoral Cutaneous Nerve Blocks for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-0063
Record Dates: First submitted 2023-06-16; First posted 2023-08-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Replacement; Genicular Nerve Block; Opioid Use
MeSH Terms: interventions — Bupivacaine; Calcium Dobesilate; Fentanyl; Mepivacaine

STUDY DESIGN:
Intervention Model Description: A randomized control trial of two groups, intervention vs. control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Once an individual enrolls, research staff will give the anesthesiologist (a co-investigator) an opaque envelope. Inside the envelope will be an index card to let them know which group the participant is assigned to (intervention or control).
  Those who will be blinded as to which group the participant is assigned to are:
  * Participant
  * Research personnel (research assistants)
  Those who will not be blinded as to which group the participant is assigned to are:
  * Primary Investigator
  * Co-investigator
  * Biostatistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 Standard TKA (No Intervention): The standard TKA group will receive the standard of care analgesia. Those in the control group will be given 7 mg of the preservative dexamethasone intravenously.
  The standard group will be given 2-5 mg of intravenous midazolam and up to 100 mcg fentanyl for sedation and analgesia while the peripheral nerve blocks and spinal anesthesia are being performed. All patients will receive a spinal anesthetic (1.5% mepivacaine 52.5 - 60mg) as well as the standard adductor canal block and infiltration between the popliteal artery and posterior knee capsule block (20 ml of 0.25% bupivacaine with 2 mg preservative free dexamethasone for each block).
- Group 2 Genicular TKA (Experimental): The genicular group will receive the study intervention of a genicular nerve block and anterior femoral cutaneous nerve block. The intervention group (genicular nerve block/anterior femoral cutaneous nerve block) will receive additional nerve blocks totaling 30 ml of 0.25% bupivacaine with 4 mg preservative-free dexamethasone (5 ml for each block: SMGN, IMGN, SLGN, NVI; 10ml for AFCN).
  The genicular group will be given 2-5 mg of intravenous midazolam and up to 100 mcg fentanyl for sedation and analgesia while the peripheral nerve blocks and spinal anesthesia are being performed. All patients will receive a spinal anesthetic (1.5% mepivacaine 52.5 - 60mg) and the standard adductor canal block and infiltration between the popliteal artery and posterior knee capsule block (20 ml of 0.25% bupivacaine with 2 mg preservative free dexamethasone for each block).
  Interventions: Drug: Bupivacaine Injection; Drug: Dexamethasone injection; Drug: Fentanyl; Drug: Mepivacaine

INTERVENTIONS:
Drug: Bupivacaine Injection — The genicular nerve block and anterior femoral cutaneous nerve blocks consists of bupivacaine with preservative-free dexamethasone injections.
  Other Names: Marcaine
  Arms: Group 2 Genicular TKA
Drug: Dexamethasone injection — The genicular nerve block and anterior femoral cutaneous nerve blocks consists of bupivacaine with preservative-free dexamethasone injections.
  Other Names: Ozurdex
  Arms: Group 2 Genicular TKA
Drug: Fentanyl — This is a drug that is given as part of the analgesia and sedation regime. This drug is not the study intervention.
  Other Names: Actiq
  Arms: Group 2 Genicular TKA
Drug: Mepivacaine — This is a drug that is given as part of the analgesia and sedation regime. This drug is not the study intervention.
  Other Names: Carbocaine
  Arms: Group 2 Genicular TKA

SUMMARY:
The goal of this randomized controlled trial is to examine if there is a relationship between the addition of the genicular nerve block and anterior femoral cutaneous nerve block in providing analgesia and the use of oral and intravenous medication in patients undergoing a total knee arthroplasty. The main questions it aims to answer are:

1. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care reduce patients' total opioid consumption in the first 24 hours after total knee arthroplasty (TKA) surgery?
2. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care reduce patients' worst numeric rating scale (NRS) pain score in the post-anesthesia care unit (PACU)?
3. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care result in earlier discharge from the post-anesthesia care unit (PACU)?
4. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care reduce patients' total opioid consumption in the first 7 days after total knee arthroplasty (TKA) surgery?
5. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care reduce patients' numerical rating scale (NRS) pain (both at rest and during movement) in the first 24 and 48 hours after surgery?

Participants will be randomly assigned to receive the genicular nerve block and anterior femoral cutaneous nerve block in addition to standard of care (intervention group), or not receive the nerve blocks (control group).

Comparing the intervention group to the control group, the researcher's primary outcomes are numerical pain in the post-anesthesia care unit and cumulative opioid consumption during the first 24 hours.

DETAILED DESCRIPTION:
Adductor canal nerve block (ACB), infiltration between the popliteal artery and the posterior knee capsule (IPACK), with or without peri-articular infiltration of local anesthetics (PAI), is the current standard of practice for analgesia coverage after total knee arthroplasty at the Hospital for Special Surgery. However, we frequently see patients with moderate post-operative knee pain, particularly on the anterior, middle, and lateral sides of the knee. There is limited clinical research on if adding a genicular nerve block could offer TKA patients a more complete analgesia. This study will test if the addition of genicular nerve block (including superolateral genicular nerve, superomedial genicular nerve, inferomedial genicular nerve, and nerve to vastus intermedius) and anterior femoral cutaneous nerve block could offer TKA patients a more complete analgesia. Participants will be randomly assigned to receive the genicular nerve block and anterior femoral cutaneous nerve block in addition to standard of care (intervention group), or not receive the nerve blocks (control group).

The main questions it aims to answer are:

1. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care reduce patients' total opioid consumption in the first 24 hours after total knee arthroplasty (TKA) surgery?
2. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care reduce patients' worst numeric rating scale (NRS) pain score in the post-anesthesia care unit (PACU)?
3. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care result in earlier discharge from the post-anesthesia care unit (PACU)?
4. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care reduce patients' total opioid consumption in the first 7 days after total knee arthroplasty (TKA) surgery?
5. Does incorporating genicular nerve block and anterior femoral cutaneous nerve block to our current standard of care reduce patients' numerical rating scale (NRS) pain (both at rest and during movement) in the first 24 and 48 hours after surgery?

Participants will be randomly assigned to receive the genicular nerve block and anterior femoral cutaneous nerve block in addition to standard of care (intervention group), or not receive the nerve blocks (control group).

Comparing the intervention group to the control group, the researcher's primary outcomes are numerical pain in the post-anesthesia care unit and cumulative opioid consumption during the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18-80
* patients undergoing ambulatory unilateral total knee arthroplasty, including 23 hour stay cohort
* ASA I-III
* BMI < 35

Exclusion Criteria:

* history of chronic pain syndromes
* chronic opioid use (daily morphine milligram equivalents > 30 mg for at least 3 months)
* contraindication to peripheral nerve blocks
* contraindication to neuraxial anesthesia
* history of peripheral neuropathy or pre-existing neurological deficits
* Psychiatrics or cognitive disorder that prohibit patient from following study protocol
* allergy to local anesthetic or study medications
* multiligament surgery
* history of substance abuse
* infection at the site of injection
* chronic kidney disease
* currently taking anticonvulsants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) pain score | in the post-operative care unit (PACU) up to 24 hours after surgery end
  The numeric rating scale (NRS) is a pain screening tool used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Cumulative opioid consumption | 24 hours after surgery end
  The cumulative opioid consumption measured in oral morphine equivalent (OME).

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) pain score | at post operative day 1 and post operative day 2
  The numeric rating scale (NRS) is a pain screening tool used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
  Although measured at different time points the average score at each time point is reported among all participants.
Cumulative opioid consumption | at post operative day 1, 2, & 7
  The cumulative opioid consumption measured in oral morphine equivalent (OME). Measured at 3 timepoints - POD 1, 2 and 7
Brief Pain Inventory (short form) | in the post-operative care unit (PACU), up to 24 hours after surgery end and at 7 days after the day of surgery
  The Brief Pain Inventory - Short Form (BPI-sf) is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. Measured on a scale from 0 to 10.
  Scoring:
  1 - 4 = Mild Pain 5 - 6 = Moderate Pain 7 - 10 = Severe Pain
  Although measured at different time points the average score at each time point is reported among all participants.
Participant satisfaction with pain treatment | in the post-operative care unit (PACU), up to 24 hours after surgery end and at 7 days after the day of surgery
  To assess patients' satisfaction with their pain management. Measured on a scale from 0 to 10, with 0 = strongly dissatisfied and 10 = strongly satisfied.
  Although measured at different time points the average score at each time point is reported among all participants.
Readiness for home discharge | from induction end (time zero) to readiness for discharge time, up to 7 days
  From time zero, the time when the patient is ready for discharge. Time zero corresponds to the time when anesthesia induction is complete (induction end). A subgroup analysis for this outcome is planned, with 1) a primary analysis of all patients discharged on the day of surgery and 2) a secondary analysis of all patients discharged 23 hours after time zero or whose status was changed to inpatient.
Bang Blinding Index | at 7 days after surgery
  To assess the success of patient and research staff blinding using the bang blinding index.
  The Bang Blinding Index is calculated per treatment arm, is a continuous value such that -1 <= Bang BI <= 1. If the index is 1, all responses are correct, and complete unblinding is inferred.

CONTACTS AND LOCATIONS:
Overall Officials: Jiabin Liu, MD/PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Conger A, Gililland J, Anderson L, Pelt CE, Peters C, McCormick ZL. Genicular Nerve Radiofrequency Ablation for the Treatment of Painful Knee Osteoarthritis: Current Evidence and Future Directions. Pain Med. 2021 Jul 25;22(Suppl 1):S20-S23. doi: 10.1093/pm/pnab129. PMID 34308957
- [Result] Kim DH, Choi SS, Yoon SH, Lee SH, Seo DK, Lee IG, Choi WJ, Shin JW. Ultrasound-Guided Genicular Nerve Block for Knee Osteoarthritis: A Double-Blind, Randomized Controlled Trial of Local Anesthetic Alone or in Combination with Corticosteroid. Pain Physician. 2018 Jan;21(1):41-52. PMID 29357330
- [Result] Rambhia M, Chen A, Kumar AH, Bullock WM, Bolognesi M, Gadsden J. Ultrasound-guided genicular nerve blocks following total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2021 Oct;46(10):862-866. doi: 10.1136/rapm-2021-102667. Epub 2021 Jul 14. PMID 34261807

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT05980546/Prot_SAP_001.pdf